CLINICAL TRIAL: NCT01535742
Title: Prospective Randomized Comparison of the Ambu Aura-i and Air-Q Intubating Laryngeal Airways as a Conduit for Tracheal Intubation in Children
Brief Title: Ambu Aura-i and Air-Q Intubating Laryngeal Airways as a Conduit for Tracheal Intubation in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Principal Investigator, Narasimhan Jagannathan, primary investigator; MD, Ann & Robert H Lurie Children's Hospital of Chicago
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: Air-Q versus Ambu-Aura-i
Record Dates: First submitted 2012-02-13; First posted 2012-02-20 (Estimated); Last update posted 2012-06-29 (Estimated); Status verified 2012-06

CONDITIONS: Tracheal Intubation in Children
Keywords: laryngeal mask airway; children; tracheal intubation; fiberoptic bronchoscopy

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (4):
- Ambu Aura-i size 1.5 (Experimental): patients will receive either the Ambu Aura-i size 1.5 or air-Q ILA 1.5 based on manufacturer recommendations of body weight
  Interventions: Device: Ambu Aura-i size 1.5
- air-Q size 1.5 (Experimental): patients will receive either the Ambu Aura-i size 1.5 or air-Q ILA 1.5 based on manufacturer recommendations of body weight
  Interventions: Device: air-Q ILA size 1.5
- Ambu Aura-i size 2 (Experimental): patients will receive either the Ambu Aura-i size 2 or air-Q ILA 2 based on manufacturer recommendations of body weight
  Interventions: Device: Ambu Aura-i size 2
- air-Q size 2 (Experimental): patients will receive either the Ambu Aura-i size 2 or air-Q ILA 2 based on manufacturer recommendations of body weight
  Interventions: Device: air-Q ILA size 2

INTERVENTIONS:
Device: Ambu Aura-i size 1.5 — Device will be placed and fiberoptic tracheal intubation will be performed and timed. Laryngeal grade of view will also be assessed
  Arms: Ambu Aura-i size 1.5
Device: air-Q ILA size 1.5 — Device will be placed and fiberoptic tracheal intubation will be performed and timed. Laryngeal grade of view will also be assessed
  Arms: air-Q size 1.5
Device: Ambu Aura-i size 2 — Device will be placed and fiberoptic tracheal intubation will be performed and timed. Laryngeal grade of view will also be assessed
  Arms: Ambu Aura-i size 2
Device: air-Q ILA size 2 — Device will be placed and fiberoptic tracheal intubation will be performed and timed. Laryngeal grade of view will also be assessed
  Arms: air-Q size 2

SUMMARY:
The purpose of this study is to determine whether there is a clinically relevant difference in time to tracheal intubation when using fiberoptic bronchoscope as a guide to intubate through the Ambu Aura-i or air-Q ILA.

DETAILED DESCRIPTION:
The goal of this prospective randomized study is to compare the Ambu Aura-i and air-Q ILA in children with normal airway anatomy, in order to evaluate the effectiveness of fiberoptic tracheal intubation through these two devices. The ease of placement, fiberoptic grade of laryngeal view, time to tracheal intubation, time for device removal after intubation, and peri-operative complications will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Children undergoing general anesthesia requiring tracheal intubation
* Weight 5-20 kg
* Age one month-six years

Exclusion Criteria:

* ASA class IV, V Emergency procedures
* History of a difficult airway
* Active upper respiratory tract infection
* Children receiving emergent surgery

Ages: 1 Month to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2012-02; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Ease and time to successful tracheal intubation | participants will be followed for the duration of anesthesia and after surgery, an expected average of 12 hours
  from the time of fiberoptic bronchoscope entry into the device until positive clinical signs indicating successful tracheal intubation (i.e., presence of bilateral breath sounds, appropriate end-tidal CO2) are confirmed

SECONDARY OUTCOMES:
Ease and time to place airway | participants will be followed for the duration of anesthesia and after surgery, an expected average of 12 hours
  From picking up the airway device to bilateral chest expansion and presence of ETCO2
Number of attempts to place the supraglottic device and tracheal tube | participants will be followed for the duration of anesthesia and after surgery, an expected average of 12 hours
  number of attempts needed for successful placement will be recorded (maximum of 3 attempts; >3 attempts will be considered as a failure)
Airway Leak Pressure | participants will be followed for the duration of anesthesia and after surgery, an expected average of 12 hours
  Airway leak pressures will be measured by recording the circuit pressure at which equilibrium is reached when fresh gas flow is delivered at 3L/min when the pressure limiting valve is closed completely
Fiberoptic grade of laryngeal view | participants will be followed for the duration of anesthesia and after surgery, an expected average of 12 hours
  The laryngeal alignment through the devices will be graded using an established scoring system
Time to remove device | participants will be followed for the duration of anesthesia and after surgery, an expected average of 12 hours
  removal will be done with the use of a removal stylet. Should inadvertent extubation occur during removal of the device, the intubation will be deemed a failure.
Airway maneuvers | participants will be followed for the duration of anesthesia and after surgery, an expected average of 12 hours
  The number and type of various airway maneuvers such as jaw thrust, neck extension, advancement/ withdrawal of the supraglottic device, and/ or anterior Laryngeal Pressure to optimize tracheal intubation will be recorded
Adverse effects | Participants will be followed for the duration of anesthesia and 24 hours postoperatively
  complications such as oxygen desaturations, inadvertent extubation, tracheal pilot balloon breakage, mucosal trauma, reflex activation of the airway, sore throat, dysphonia will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Narasimhan Jagannathan, MD, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (1):
- Childrens Memorial Hospital, Chicago, Illinois, United States

REFERENCES:
- [Background] Jagannathan N, Sohn LE, Mankoo R, Langen KE, Mandler T. A randomized crossover comparison between the Laryngeal Mask Airway-Unique and the air-Q intubating laryngeal airway in children. Paediatr Anaesth. 2012 Feb;22(2):161-7. doi: 10.1111/j.1460-9592.2011.03703.x. Epub 2011 Sep 15. PMID 21917058
- [Background] Jagannathan N, Kozlowski RJ, Sohn LE, Langen KE, Roth AG, Mukherji II, Kho MF, Suresh S. A clinical evaluation of the intubating laryngeal airway as a conduit for tracheal intubation in children. Anesth Analg. 2011 Jan;112(1):176-82. doi: 10.1213/ANE.0b013e3181fe0408. Epub 2010 Nov 16. PMID 21081777
- [Background] Sinha R, Chandralekha, Ray BR. Evaluation of air-Q intubating laryngeal airway as a conduit for tracheal intubation in infants--a pilot study. Paediatr Anaesth. 2012 Feb;22(2):156-60. doi: 10.1111/j.1460-9592.2011.03710.x. PMID 21973052
- [Background] Baker PA, Brunette KE, Byrnes CA, Thompson JM. A prospective randomized trial comparing supraglottic airways for flexible bronchoscopy in children. Paediatr Anaesth. 2010 Sep;20(9):831-8. doi: 10.1111/j.1460-9592.2010.03362.x. PMID 20716075